CLINICAL TRIAL: NCT06519149
Title: Safety and Effectiveness of Slow Wave Device for the Treatment of Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Slow Wave, Inc. (Industry)
Collaborators: St. David's HealthCare (Other)
Responsible Party: Sponsor
Other Study IDs: 2192249-1
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Slow Wave UASD: Participants who wear the Slow Wave UASD oral device fora 90 day period and a Wellue O2 ring to measure daily sleep metrics
  Interventions: Device: Slow Wave UASD

INTERVENTIONS:
Device: Slow Wave UASD — An oral appliance for the treatment of OSA and snoring
  Other Names: Slow Wave Oral appliance for the treatment of OSA

SUMMARY:
This is a safety and efficacy trial for a Slow Wave, Inc. UASD oral appliance for the treatment of Obstructive Sleep Apnea. This trial will recruit 60-80 participants through our IRB partner. Each participant will take pre-trial and post trail sleep studies and be measured before, throughout and after the trial for Apnea-Hypopnea Index (AHI), Oxygen Desaturation Index (ODI), pulse rate to determine level of sleep improvement while wearing the device. Safety will also be measured through survey, dental exams and adverse events monitoring. Patients will wear an O2 monitoring ring throughout the study and upload results daily. Primary Objectives will evaluate AHI and ODI between sleep studies. Secondary outcomes will compare the daily ring data to these two sleep studies to evaluate changes over time. Patients will have the opportunity to complete daily diaries on their sleep experiences.

DETAILED DESCRIPTION:
This study is a single-center, single-arm open label study to evaluate the safety and effectiveness of the Slow Wave UASD sleep and snore device in individuals with mild-to-moderate Obstructive Sleep Apnea (OSA) and individuals with severe OSA of less than 40 AHI events per hour who are not able to tolerate CPAP treatment.

All participants will be given and initial Home Sleep Apnea Test (HSAT) to establish baseline readings for: Number of OSA events during sleep, average O2 score during sleep, average pulse rate and Oxygen desaturation events of more than 4% during sleep (ODI). The initial HSAT will also determine if the patients have OSA.

All participants will get an intraoral scan with a closed bite by a study partner. The 3D scan will be used to create a personalized Slow Wave UASD device that will be used throughout the study. Each participant will wear the device for a 90-day period. Each participant will be given a WellUE O2 ring to wear every night throughout the study. The ring connects to the WellUE application that participants will be asked to download to their phones. The O2 ring application collects much of hte same data as is collected in a home sleep study. Participants will be asked to upload the ring results to a study-managed database on a daily basis. Ring results will be presented as secondary objectives in this trial. The failure of a participant to send ring data will not disqualify them from the trial as primary objectives are the comparison of beginning and ending HSAT results. Patients will be given patient health questionnaires and physical examinations prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* • Provision of signed and dated informed consent form

  * Unable to tolerate or decline positive airway pressure therapy
  * Absence of markedly enlarged tonsils, defined as 3+ or 4+ according to the Brodsky classification
  * Able to protrude tongue ≥20mm beyond maxillary incisors
  * No uncontrolled nasal obstruction (must be able to breathe through nose)
  * Stable medication regimen for ≥1 month
  * Stated willingness to comply with all study procedures and availability for the duration of the study
  * Male or female, of any race, aged 18-70 years (inclusive)
  * If diagnosed with uncomplicated Mild to moderate, moderate to severe OSA (i.e., AHI >5, <30 h-1); where uncomplicated is defined by the absence of:

    * Conditions that place the patient at increased risk of non-obstructive sleep-disordered breathing (e.g., central sleep apnea, hypoventilation, and sleep-related hypoxemia). Examples of such conditions include significant cardiopulmonary disease, potential respiratory muscles weakness due to neuromuscular conditions, history of stroke, and chronic opiate medication use.
    * Concern for significant non-respiratory sleep disorder(s) that require evaluation (e.g., disorders of central hypersomnolence, parasomnias, sleep-related movement disorders) or interfere with accuracy of HSAT (e.g., severe insomnia).
    * Environmental or personal factors that preclude the adequate acquisition and interpretation of data from HSAT.
  * Body mass index (BMI) < 35 kg/m2
  * Neck circumference < 45 cm
  * Absence of severe oxyhemoglobin desaturation during sleep, indicated by mean nocturnal SpO2 > 82%
  * Mandibular range of motion > 5 mm in protrusive direction
  * Adequate dentition, as determined by the site dentist
  * Must have a smart phone able to download 02 ring app

Exclusion Criteria:

* • Inability to breathe through the nose comfortably

  * Presence of > 25% Central Sleep Apnea (CSA)
  * Severe OSA above AHI >40
  * Uncontrolled sleep disorder such as narcolepsy, chronic insomnia, restless legs syndrome, or REM behavior disorder
  * Presence of positional obstructive sleep apnea per Cartwright's definition (Ratio of respiratory events in the supine to nonsupine position greater than 2:1)
  * History of surgery intended to alter anatomy for the correction of OSA, such as uvulopalatopharyngoplasty (UPPP), maxillomandibular advancement (MMA), or tongue/hyoid suspension.
  * History of surgery intended to restore normal anatomy, such as tonsillectomy, adenoidectomy, septoplasty, or polypectomy within the previous 6 months
  * Presence of hypoglossal nerve stimulation device
  * Use of CPAP or OAT within the two weeks prior to the screening HSAT
  * Anticipated change in medical therapy during the study protocol that could alter OSA severity (e.g., weight loss surgeries; UPPP, MMA, tongue/hyoid suspension)
  * Loose teeth or advanced periodontal disease
  * Teeth extractions/Presence of a dental post implanted less than 12 months
  * Removable dentures
  * History of temporomandibular joint disorder (TMJ)
  * Resistant hypertension, defined as inadequately controlled blood pressure despite therapy with ≥ 3 oral hypertensive agents
  * Presence of congestive heart failure (NYHA Class IV), persistent/permanent atrial fibrillation, or acute coronary artery disease (STEMI/NSTEMI/USA) in the past 30 days.
  * Presence of neuromuscular diseases e.g. myasthenia gravis, amyotrophic lateral sclerosis, Guillain-Barré syndrome and muscular dystrophy, or hypoventilation disorders which results in shallow breathing during sleep and/or cyanosis of the fingers/toes.
  * Presence of pulmonary disease resulting in significant desaturation, e.g., severe chronic obstructive pulmonary disease, interstitial lung disease (SaO2 nadir of 87%), or pulmonary hypertension
  * History of cerebrovascular incident within the last 12 months
  * Use of pacemaker or other life supporting device
  * Anticipated change in body weight > 5% during the study period
  * Participation in other studies that could interfere with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with mild-to-moderate OSA and individuals with severe OSA below and AHI of 40 who cannot tolerate CPAP treatment
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
AHI Events per hour | 90 days
  A 50% or greater reduction in apnea-hypopnea index (AHI) events from the baseline reading while wearing the device
Oxygen Desaturation events during sleep | 90 days
  a 25% or greater decrease in events where oxygen desaturation is greater than or equal to 4% during sleep while wearing the device
Device safety and comfort | 90 days
  All reported adverse events and patient input of side effects, dental exams and surveys

SECONDARY OUTCOMES:
Efficacy Ring Comparison | 90 days
  comparing baseline and ending HSAT sleep study results to collected patient ring data
Pulse rate | 90 days
  effect on pulse rate while wearing the appliance
Device safety and comfort | 120 days
  development of adverse events and development of any side effects over time.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Jepson, MD, Principal Investigator — St. David's HealthCare; Nirman Koladia, MD, Study Director — Clinical Research Consultant
Locations (1):
- Austin Heart Research, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Varghese L, Rebekah G, N P, Oliver A, Kurien R. Oxygen desaturation index as alternative parameter in screening patients with severe obstructive sleep apnea. Sleep Sci. 2022 Jan-Mar;15(Spec 1):224-228. doi: 10.5935/1984-0063.20200119. PMID 35273770
- [Result] Temirbekov D, Gunes S, Yazici ZM, Sayin I. The Ignored Parameter in the Diagnosis of Obstructive Sleep Apnea Syndrome: The Oxygen Desaturation Index. Turk Arch Otorhinolaryngol. 2018 Mar;56(1):1-6. doi: 10.5152/tao.2018.3025. Epub 2018 Mar 1. PMID 29988275
- [Result] Cartwright RD. Effect of sleep position on sleep apnea severity. Sleep. 1984;7(2):110-4. doi: 10.1093/sleep/7.2.110. PMID 6740055
- See also: Market sizing information on OSA — http://www.cms.gov/medicare/coverage/evidence/cpap